CLINICAL TRIAL: NCT01807234
Title: Comparison of Ketorolac Nasal Spray to Sumatriptan Nasal Spray and Placebo for Acute Treatment of Migraine (The KSPN Migraine Study)
Brief Title: Comparison of Ketorolac Nasal Spray to Sumatriptan Nasal Spray and Placebo for Acute Treatment of Migraine
Acronym: KSPN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Regent, Inc. (Industry)
Responsible Party: Principal Investigator, Drs Barbara Peterlin, Director, The Johns Hopkins Bayview Headache Research, Johns Hopkins University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NA00075486
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Migraines
MeSH Terms: conditions — Migraine Disorders | interventions — Ketorolac; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketorolac/Placebo (Experimental): Ketorolac 31.5 mg single dose nasal spray and Placebo
  Interventions: Drug: Ketorolac; Drug: Placebo
- Sumatriptan/Placebo (Experimental): Sumatriptan 20 mg single dose nasal spray and placebo
  Interventions: Drug: Sumatriptan; Drug: Placebo
- Ketorolac Placebo/Sumatriptan placebo (Placebo Comparator): single dose Ketorolac placebo, single dose Sumatriptan placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac — Single dose of Ketorolac (Sprix) nasal spray 31.5 mg, one spray in each nostril for an acute migraine attack.
  Other Names: Sprix
  Arms: Ketorolac/Placebo
Drug: Sumatriptan — Sumatriptan (Imitrex) 20 mg one single dose of nasal spray for an acute migraine attack.
  Other Names: Imitrex
  Arms: Sumatriptan/Placebo
Drug: Placebo — Placebo one spray in each nostril and placebo one nasal spray.

SUMMARY:
The investigators propose to test the efficacy of ketorolac nasal spray versus sumatriptan nasal spray versus placebo for acute abortive therapy of migraine head pain as well as for migraine associated symptoms including nausea and allodynia.

DETAILED DESCRIPTION:
Participants are randomized to Ketorolac NS 31.5 mg, Sumatriptan NS 20 mg or placebo to treat three moderate to severe migraine attacks and switched treatments with each attack so that they received each treatment only once.

For each treated attack (moderate to severe migraine attack), participants utilized two study treatments (A and B). Study treatment A administered as one spray in each nostril, and study treatment B administered as one spray in one nostril.

Randomized to Ketorolac, A=Ketorolac, B=Placebo Randomized to Sumatriptan, A=Placebo, B=Sumatriptan Randomized to Placebo, A=Placebo, B=Placebo

ELIGIBILITY:
Inclusion/Exclusion Criteria

At the Screening Visit, a subject must meet the following criteria to participate in this study:

1.18-65 years of age 2.Fulfills International Classification of Headache Disorders (ICHD)-II Criteria of migraine as noted below in Table 1 3.History of migraines for at least one year 4.Migraine onset prior to the age of 50 years of age 5.Headache frequency (of any headaches, migraine or non-migraine) < 9 days per month 6.At visit 2, participants must report two or more headache days during the 28-day run-in period on the headache diary. 7.At least 48 hours of freedom from headache between treated migraine attacks. 8.If currently using headache preventive medications, must be on a stable dose for at least 3 months prior to enrollment and throughout the study period and be on no more than one prophylactic agent. 9.Able to complete all study procedures, including the questionnaire (assessing demographics, headache characteristics, headache comorbidities and medical history at the initial visit and headache characteristics) and the required headache calendars, and all study visits; 10.Able to understand, read and sign an informed consent (English).

Exclusion Criteria:

1. Any condition (history or presence of) which contraindicates the use of triptans or NSAIDs including:

   * Known hypersensitivity or intolerance to triptans or NSAIDs
   * Contraindications to triptan use (uncontrolled hypertension, ischemic heart disease, prinz-metal angina, cardiac arrhythmias, multiple risk factors for atherosclerotic vascular disease, primary vasculopathies, and basilar and hemiplegic migraine)
   * Cerebrovascular disease except for mild non-specific white matter disease
   * Peripheral vascular disease or any other ischemic disease including myocardial infarction
   * Uncontrolled hypertension (systolic BP 160 mmHg or diastolic BP 95 mmHg or (both)
   * Migraine aura fulfilling ICHD-II criteria for hemiplegic or basilar-type migraine
   * Any history of chronic renal or hepatic impairment
   * Use of an ergotamine-containing medication or monamine oxidase inhibitor
   * Known or suspected pregnancy, negative pregnancy test
   * Lactation
   * Bleeding dsycrasias including gastritis, peptic ulcer disease,gastrointestinal bleeding
2. Physician diagnosis of any pain syndrome other than migraine
3. Classification as treatment resistant by investigator
4. Known drug or substance abuse
5. Any opioid use in past 2 months
6. Use of any medication, which could interfere with study assessments
7. History of noncompliance with taking medication;
8. Use of any experimental drug or device within 30 days prior to the Screening Visit (Visit 1);
9. Any abnormal finding or condition deemed clinically significant by the investigator on history, screening, or physical exam that contraindicates the use of triptans or NSAIDs or that might interfere with the patient's safety, study participation, or which might confound the interpretation of the study results.
10. Any history of chronic renal or hepatic disease already excluded above under number 1; plus see exclusion 9.
11. History of chronic pulmonary disorder including nasal polyps (see 1) and asthma.
12. History of upper respiratory infection or other respiratory tract condition that could interfere with the absorption of the nasal spray or with assessment of AEs including rhinitis medicamentosa (chronic daily use of topical decongestants).
13. History of nasal surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Johns Hopkins Bayview Headache Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rao AS, Gelaye B, Kurth T, Dash PD, Nitchie H, Peterlin BL. A Randomized Trial of Ketorolac vs. Sumatripan vs. Placebo Nasal Spray (KSPN) for Acute Migraine. Headache. 2016 Feb;56(2):331-40. doi: 10.1111/head.12767. Epub 2016 Feb 3. PMID 26840902

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketorolac Then Sumatriptan Then Placebo: Participants were randomized for three attacks. For each treated attack, participants utilized two study treatments (A and B). Study treatment A administered as one spray in each nostril, and study treatment B administered as one spray in one nostril.
  Randomized to Ketorolac, A=Ketorolac, B=Placebo Randomized to Sumatriptan, A=Placebo, B=Sumatriptan Randomized to Placebo, A=Placebo, B=Placebo
  Attack 1: Ketorolac: Single dose of Ketorolac spray 31.5 kg, one spray in each nostril for acute migraine attack (Treatment A), placebo spray (Treatment B) in one nostril.
  Attack 2: Sumatriptan: Placebo spray (treatment A) in one nostril, 20 mg single dose of Sumatriptan spray (Treatment B) into one nostril.
  Attack 3: Placebo: Placebo spray (Treatment A) in each nostril, Placebo Spray (Treatment B) in each nostril.
- Kerorolac Then Placebo Then Sumatriptan: Participants were randomized for three attacks. For each treated attack, participants utilized two study treatments (A and B). Study treatment A administered as one spray in each nostril, and study treatment B administered as one spray in one nostril.
  Randomized to Ketorolac, A=Ketorolac, B=Placebo Randomized to Sumatriptan, A=Placebo, B=Sumatriptan Randomized to Placebo, A=Placebo, B=Placebo
  Attack 1: Ketorolac: Single dose of Ketorolac spray 31.5 kg, one spray in each nostril for acute migraine attack (Treatment A), placebo spray (Treatment B) in one nostril.
  Attack 2: Placebo: Placebo spray (Treatment A) in each nostril, Placebo Spray (Treatment B) in each nostril.
  Attack 3: Sumatriptan: Placebo spray (treatment A) in one nostril, 20 mg single dose of Sumatriptan spray (Treatment B) into one nostril.
- Sumatriptan Then Ketorolac Then Placebo: Participants were randomized for three attacks. For each treated attack, participants utilized two study treatments (A and B). Study treatment A administered as one spray in each nostril, and study treatment B administered as one spray in one nostril.
  Randomized to Ketorolac, A=Ketorolac, B=Placebo Randomized to Sumatriptan, A=Placebo, B=Sumatriptan Randomized to Placebo, A=Placebo, B=Placebo
  Attack 1: Sumatriptan: Placebo spray (treatment A) in one nostril, 20 mg single dose of Sumatriptan spray (Treatment B) into one nostril.
  Attack 2: Ketorolac: Single dose of Ketorolac spray 31.5 kg, one spray in each nostril for acute migraine attack (Treatment A), placebo spray (Treatment B) in one nostril.
  Attack 3: Placebo: Placebo spray (Treatment A) in each nostril, Placebo Spray (Treatment B) in each nostril.
- Sumatriptan Then Placebo Then Ketorolac: Participants were randomized for three attacks. For each treated attack, participants utilized two study treatments (A and B). Study treatment A administered as one spray in each nostril, and study treatment B administered as one spray in one nostril.
  Randomized to Ketorolac, A=Ketorolac, B=Placebo Randomized to Sumatriptan, A=Placebo, B=Sumatriptan Randomized to Placebo, A=Placebo, B=Placebo
  Attack 1: Sumatriptan: Placebo spray (treatment A) in one nostril, 20 mg single dose of Sumatriptan spray (Treatment B) into one nostril.
  Attack 2: Placebo: Placebo spray (Treatment A) in each nostril, Placebo Spray (Treatment B) in each nostril.
  Attack 3: Ketorolac: Single dose of Ketorolac spray 31.5 kg, one spray in each nostril for acute migraine attack (Treatment A), placebo spray (Treatment B) in one nostril.
- Placebo Then Ketorolac Then Sumatriptan: Participants were randomized for three attacks. For each treated attack, participants utilized two study treatments (A and B). Study treatment A administered as one spray in each nostril, and study treatment B administered as one spray in one nostril.
  Randomized to Ketorolac, A=Ketorolac, B=Placebo Randomized to Sumatriptan, A=Placebo, B=Sumatriptan Randomized to Placebo, A=Placebo, B=Placebo
  Attack 1: Placebo: Placebo spray (Treatment A) in each nostril, Placebo Spray (Treatment B) in each nostril.
  Attack 2: Ketorolac: Single dose of Ketorolac spray 31.5 kg, one spray in each nostril for acute migraine attack (Treatment A), placebo spray (Treatment B) in one nostril.
  Attack 3: Sumatriptan: Placebo spray (treatment A) in one nostril, 20 mg single dose of Sumatriptan spray (Treatment B) into one nostril.
- Placebo Then Sumatriptan Then Ketorolac: Participants were randomized for three attacks. For each treated attack, participants utilized two study treatments (A and B). Study treatment A administered as one spray in each nostril, and study treatment B administered as one spray in one nostril.
  Randomized to Ketorolac, A=Ketorolac, B=Placebo Randomized to Sumatriptan, A=Placebo, B=Sumatriptan Randomized to Placebo, A=Placebo, B=Placebo
  Attack 1: Placebo: Placebo spray (Treatment A) in each nostril, Placebo Spray (Treatment B) in each nostril.
  Attack 2: Sumatriptan: Placebo spray (treatment A) in one nostril, 20 mg single dose of Sumatriptan spray (Treatment B) into one nostril.
  Attack 3: Ketorolac: Single dose of Ketorolac spray 31.5 kg, one spray in each nostril for acute migraine attack (Treatment A), placebo spray (Treatment B) in one nostril.
Period: Overall Study
Arm/Group | Ketorolac Then Sumatriptan Then Placebo | Kerorolac Then Placebo Then Sumatriptan | Sumatriptan Then Ketorolac Then Placebo | Sumatriptan Then Placebo Then Ketorolac | Placebo Then Ketorolac Then Sumatriptan | Placebo Then Sumatriptan Then Ketorolac
Started | 12 | 12 | 12 | 12 | 12 | 12
Randomized, But Did Not Take Drug | 3 | 5 | 2 | 1 | 4 | 3
Completed Only 1 Attack | 2 | 1 | 0 | 1 | 0 | 1
Completed | 7 | 6 | 10 | 10 | 8 | 8
Not Completed | 5 | 6 | 2 | 2 | 4 | 4
Not completed — Lost to Follow-up | 2 | 5 | 1 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 1 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Of the 72 randomized participants, 54 (75%) treated at least one attack and 49 (68%) completed all three treatments, for a total of 152 treated migraine attacks.
Groups:
- Ketorolac Then Placebo Then Sumatriptan: Participants were randomized for three attacks. For each treated attack, participants utilized two study treatments (A and B). Study treatment A administered as one spray in each nostril, and study treatment B administered as one spray in one nostril.
  Randomized to Ketorolac, A=Ketorolac, B=Placebo Randomized to Sumatriptan, A=Placebo, B=Sumatriptan Randomized to Placebo, A=Placebo, B=Placebo
  Attack 1: Ketorolac: Single dose of Ketorolac spray 31.5 kg, one spray in each nostril for acute migraine attack (Treatment A), placebo spray (Treatment B) in one nostril.
  Attack 2: Placebo: Placebo spray (Treatment A) in each nostril, Placebo Spray (Treatment B) in each nostril.
  Attack 3: Sumatriptan: Placebo spray (treatment A) in one nostril, 20 mg single dose of Sumatriptan spray (Treatment B) into one nostril.
- Total: Total of all reporting groups
Arm/Group | Ketorolac Then Sumatriptan Then Placebo | Ketorolac Then Placebo Then Sumatriptan | Sumatriptan Then Ketorolac Then Placebo | Sumatriptan Then Placebo Then Ketorolac | Placebo Then Ketorolac Then Sumatriptan | Placebo Then Sumatriptan Then Ketorolac | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 12 | 12 | 12 | 12 | 72
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Average age of participants
  years | 36.3 (9.8) | 36.3 (9.8) | 36.3 (9.8) | 36.3 (9.8) | 36.3 (9.8) | 36.3 (9.8) | 36.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 12 | 12 | 12 | 11 | 70
  Male | 1 | 0 | 0 | 0 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 12 | 12 | 12 | 72

OUTCOME MEASURES:

1. Primary Outcome: 2- Hour Pain Relief
Description: The primary outcome was 2-hour headache relief; headache relief was defined as headache pain from moderate or severe pain to none or mild pain. Pain was assessed using a 4-point scale (none, mild, moderate, and severe)
Time Frame: 2 hours
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ketorolac/ Placebo: Ketorolac 31.5 mg single dose nasal spray and Placebo
  Ketorolac: Single dose of Ketorolac nasal spray 31.5 mg, one spray in each nostril for an acute migraine attack.
  Placebo: Ketorolac placebo one spray in each nostril and Sumatriptan placebo one nasal spray.
- Sumatriptan/ Placebo: Sumatriptan 20 mg single dose nasal spray and placebo
  Sumatriptan: Sumatriptan 20 mg one single dose of nasal spray for an acute migraine attack.
  Placebo: SPRIX placebo one spray in each nostril and Sumatriptan placebo one nasal spray.
- Ketorolac Placebo/ Sumatriptan Placebo: Single dose Ketorolac placebo, single dose Sumatriptan placebo
  Placebo: Ketorolac placebo one spray in each nostril and Sumatriptan placebo one nasal spray.
Arm/Group | Ketorolac/ Placebo | Sumatriptan/ Placebo | Ketorolac Placebo/ Sumatriptan Placebo
Number analyzed (Participants) | 52 | 50 | 50
percentage of participants | 72.5 [59.9 to 85.2] | 69.4 [56.0 to 82.8] | 38.8 [24.6 to 52.9]

2. Secondary Outcome: Pain Freedom
Description: 1) Pain Freedom: Pain Freedom at 2 hours is defined as being free of pain. Pain was assessed using a 4-point scale (none, mild, moderate, and severe).
Time Frame: 2-hours
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Sumatriptan/Placebo: Sumatriptan 20 mg single dose nasal spray and placebo
  Sumatriptan: Sumatriptan 20 mg one single dose of nasal spray for an acute migraine attack.
  Placebo: Ketorolac placebo one spray in each nostril and Sumatriptan placebo one nasal spray.
Arm/Group | Ketorolac/ Placebo | Sumatriptan/Placebo | Ketorolac Placebo/ Sumatriptan Placebo
Number analyzed (Participants) | 52 | 50 | 50
percentage of patients | 43.1 [29.1 to 57.2] | 36.7 [22.7 to 50.7] | 18.4 [7.1 to 29.6]

3. Secondary Outcome: Absence of Photophobia
Description: 2) Defined as reduction of photophobia to none. Symptom was assessed using a 4-point scale (none, mild, moderate, and severe)
Time Frame: 2-hours
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Sumatriptan/ Placebo: Sumatriptan 20 mg single dose nasal spray and placebo
  Sumatriptan: Sumatriptan 20 mg one single dose of nasal spray for an acute migraine attack.
  Placebo: Ketorolac placebo one spray in each nostril and Sumatriptan placebo one nasal spray.
Arm/Group | Ketorolac/ Placebo | Sumatriptan/ Placebo | Ketorolac Placebo/ Sumatriptan Placebo
Number analyzed (Participants) | 52 | 50 | 50
percentage of patients | 65.4 [56.1 to 74.7] | 64.0 [54.4 to 73.6] | 46.0 [36.1 to 55.9]

4. Secondary Outcome: Absence of Phonophobia
Description: 3) Defined as reduction of phonophobia to none. Symptom was assessed using a 4-point scale (none, mild, moderate, and severe)
Time Frame: 2-hours
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Ketorolac/ Placebo | Sumatriptan/Placebo | Ketorolac Placebo/ Sumatriptan Placebo
Number analyzed (Participants) | 52 | 50 | 50
percentage of patients | 75.0 [66.5 to 83.4] | 66.0 [56.5 to 75.4] | 56.0 [46.1 to 65.9]

5. Secondary Outcome: Absence of Nausea
Description: 4) Defined as reduction of nausea to none. Symptom was assessed using a 4-point scale (none, mild, moderate, and severe)
Time Frame: 2-hours
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Ketorolac/ Placebo | Sumatriptan/ Placebo | Ketorolac Placebo/ Sumatriptan Placebo
Number analyzed (Participants) | 52 | 50 | 50
percentage of patients | 82.7 [75.3 to 90.0] | 74.0 [65.2 to 82.7] | 66.0 [56.5 to 75.4]

6. Secondary Outcome: Absence of Allodynia
Description: 5) Absence of allodynia The presence of allodynia was assessed based on a series of 8 questions inquiring as to the presence of allodynia. Participants answering 2 or more questions positively were considered to have allodynia.
Time Frame: 2-hours
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Ketorolac/ Placebo | Sumatriptan/ Placebo | Ketorolac Placebo/ Sumatriptan Placebo
Number analyzed (Participants) | 52 | 50 | 50
percentage of patients | 70.5 [57.6 to 83.5] | 75.5 [63.0 to 87.9] | 69.0 [57.6 to 83.5]

7. Secondary Outcome: Self-assessment of Disability: Percentage of Participants With Moderate or Severe Disability
Description: Participants' self-assessment of disability was assessed using 4-point scales (none, mild, moderate, and severe). A binary outcome variable was created grouping none and mild vs moderate to severe. .
Time Frame: 2-hours
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Ketorolac/ Placebo | Sumatriptan/ Placebo | Ketorolac Placebo/ Sumatriptan Placebo
Number analyzed (Participants) | 52 | 50 | 50
percentage of patients | 1.9 [0.2 to 13.1] | 8.1 [3.0 to 20.1] | 10.2 [4.2 to 22.5]

8. Secondary Outcome: Sustained Pain Relief (SPR)
Description: 7) 24 and 48 hours sustained pain relief (SPR) Defined as the reduction of pain to none or mild from moderate or severe, on a 4-point scale (none, mild, moderate, and severe).
Time Frame: 24 and 48 hours
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Ketorolac/ Placebo | Sumatriptan/ Placebo | Ketorolac Placebo/ Sumatriptan Placebo
Number analyzed (Participants) | 52 | 50 | 50
percentage of patients
  24 hour sustained pain relief | 49.0 [34.8 to 63.2] | 40.8 [26.5 to 55.1] | 20.4 [8.7 to 32.1]
  48 hour sustained pain relief | 49.0 [34.8 to 63.2] | 30.6 [17.2 to 43.9] | 20.4 [8.7 to 32.1]

9. Secondary Outcome: Sustained Pain Freedom (SPF)
Description: 8) 24 and 48 hours sustained pain freedom (SPF); Defined as the reduction of pain to none. Pain was assessed using a 4-point scale (none, mild, moderate, and severe).
Time Frame: 24 and 48 hours
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Ketorolac/ Placebo | Sumatriptan/ Placebo | Ketorolac Placebo/ Sumatriptan Placebo
Number analyzed (Participants) | 52 | 50 | 50
percentage of patients
  24 hour sustained pain freedom | 35.3 [21.7 to 48.9] | 22.4 [10.3 to 34.5] | 12.2 [2.7 to 21.7]
  48 hour sustained pain freedom | 33.3 [19.9 to 46.7] | 18.4 [7.1 to 29.6] | 12.2 [2.7 to 21.7]

10. Secondary Outcome: Time to Pain Relief
Description: 9) The time, in minutes, will be measured from the time study drug is taken to the time when significant pain relief is first observed and maintained through 2 hours with no rescue medication use at or prior to this point.
Time Frame: following each treated migraine attack
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Ketorolac/ Placebo | Sumatriptan/ Placebo | Ketorolac Placebo/ Sumatriptan Placebo
Number analyzed (Participants) | 52 | 50 | 50
percentage of patients
  10 minutes | 15.7 [5.3 to 26.0] | 14.3 [4.1 to 24.4] | 12.2 [2.7 to 21.7]
  15 minutes | 35.3 [21.7 to 48.8] | 36.0 [22.2 to 49.7] | 14.3 [4.1 to 24.4]
  20 minutes | 43.1 [29.1 to 57.2] | 44.9 [30.4 to 59.3] | 22.4 [10.3 to 34.5]
  30 minutes | 54.9 [40.7 to 69.0] | 53.1 [38.6 to 67.5] | 26.5 [13.7 to 39.3]
  1 hour | 58.8 [44.8 to 72.8] | 57.1 [42.8 to 71.5] | 32.6 [19.0 to 46.2]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at the 10 minute, 15 minute, 20 minute, 30 minute, 60 minute, 2 hour, 24 hour and 72 hour mark.
Description: At each of the time intervals listed above, participants were instructed to document any adverse effects from drug that occured.
Groups:
- Sprix/Placebo: Sprix 31.5 mg single dose nasal spray and Placebo
  SPRIX: Single dose of Sprix nasal spray 31.5 mg, one spray in each nostril for an acute migraine attack.
  Placebo: SPRIX placebo one spray in each nostril and Sumatriptan placebo one nasal spray.
  The most common adverse events reported by participants treated with ketorolac NS were burning of nose, (mild in 25.5%, moderate in 19.6% and severe in 3.9%), unusual taste (mild in 2%, moderate in 5.9%, severe 2%), nasal discomfort (8%), burning of throat (6%), fatigue (4%), dizziness (4%), nausea (2%), rash (2%).
- Sumatriptan/Placebo: Sumatriptan 20 mg single dose nasal spray and placebo
  Sumatriptan: Sumatriptan 20 mg one single dose of nasal spray for an acute migraine attack.
  Placebo: SPRIX placebo one spray in each nostril and Sumatriptan placebo one nasal spray.
  For those treated with sumatriptan NS the most common adverse events were unusual taste (mild in 24.5%, moderate in 12.2%, severe 4.1%), burning of the nose (mild in 6.1%, moderate in 2%), nausea (8%), burning of the throat (6%), nasal discomfort (6%), dizziness (4%), fatigue (4%) and rash (2%).
- SRIX Placebo/Sumatriptan Placebo: single dose SPRIX placebo, single dose Sumatriptan placebo
  Placebo: SPRIX placebo one spray in each nostril and Sumatriptan placebo one nasal spray.
  The most common adverse event for placebo were unusual taste (mild in 4%, moderate in 2%), nausea (4%), rash (4%), fatigue (4%), burning of the nose (2%), dizziness (2%).
Arm/Group | Sprix/Placebo | Sumatriptan/Placebo | SRIX Placebo/Sumatriptan Placebo
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 43/52 | 39/50 | 11/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sprix/Placebo (N=52) | Sumatriptan/Placebo (N=50) | SRIX Placebo/Sumatriptan Placebo (N=50)
mild burning of nose (Respiratory, thoracic and mediastinal disorders) | 13 | 3 | 1
moderate burning of nose (Respiratory, thoracic and mediastinal disorders) | 10 | 1 | 0
severe burning of nose (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
mild unusual taste (Nervous system disorders) | 1 | 12 | 2
moderate unusual taste (Nervous system disorders) | 3 | 6 | 1
severe unusual taste (Nervous system disorders) | 1 | 2 | 0
nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0
burning of throat (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0
fatigue (General disorders) | 2 | 2 | 2
dizziness (Nervous system disorders) | 2 | 2 | 1
nausea (Gastrointestinal disorders) | 1 | 4 | 2
rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2

LIMITATIONS AND CAVEATS:
Small study size (n=54)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No